CLINICAL TRIAL: NCT04382755
Title: A Prospective Randomized Open-label Interventional Study to Investigate the Efficacy of Complement C5 Inhibition With Zilucoplan® in Improving Oxygenation and Short-and Longterm Outcome of COVID19 Patients With Acute Hypoxic Respiratory Failure
Brief Title: Zilucoplan® in Improving Oxygenation, Short-, Longterm Outcome of COVID19 Patients With Acute Hypoxic Respiratory Failure
Acronym: ZILU-COV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Bart N. Lambrecht, Professor in Pulmonology, Director VIB-Inflammational Research Center, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZILU-COV
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: Acute Lung Injury; Hypoxia; Corona virus; COVID-19; SARS (Severe Acute Respiratory Syndrome); Acute Respiratory Distress Syndrome; ARDS
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Hypoxia; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (active) (Active Comparator): Standard of Care (SoC) + subcutaneous Zilucoplan® + prophylactic antibiotics until 14 days after last Zilucoplan®
  Interventions: Drug: Zilucoplan®
- Group B (control) (Placebo Comparator): Standard of Care (SoC) + 1 week of prophylactic antibiotics (or until hospital discharge, whichever comes first)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zilucoplan® — 14 days of SC Zilucoplan® on top of standard of care + prophylactic antibiotics until 14 days after last Zilucoplan®
  Arms: Group A (active)
Drug: Placebo — standard of care treatment + 1 week of prophylactic antibiotics (or until hospital discharge, whichever comes first)
  Arms: Group B (control)

SUMMARY:
The study is a randomized controlled, open-label trial comparing subcutaneous Zilucoplan® with standard of care to standard of care alone.

In the active group, Zilucoplan® will be administered subcutaneously once daily for 14 days or till discharge from the hospital, whichever comes first.

The hypothesis of the proposed intervention is that Zilucoplan® (complement C5 inhibitor) has profound effects on inhibiting acute lung injury post COVID-19, and can promote lung repair mechanisms, that lead to a 25% improvement in lung oxygenation parameters. This hypothesis is based on experiments performed in mice showing that C5a blockade can prevent mortality and prevent ARDS in mice with post-viral acute lung injury.

Eligible patients include patients with confirmed COVID-19 infection suffering from hypoxic respiratory failure defined as O2 saturation below 93% on minimal 2l/min O2 therapy and/or ratio PaO2/FiO2 below 350.

DETAILED DESCRIPTION:
This investigator-initiated trial is a phase 2 academic, prospective, 2:1 randomized, open-label, multicenter interventional study designed to investigate the efficacy of subcutaneous Zilucoplan® in improving oxygenation and short- and long-term outcome of COVID-19 patients with acute hypoxic respiratory failure. The hypothesis of the proposed intervention is that Zilucoplan® has profound effects on inhibiting acute lung injury induced by COVID-19, and can promote lung repair mechanisms, that lead to a 25% improvement in lung oxygenation parameters. This hypothesis is based on experiments performed in mice showing that C5a blockade can prevent mortality and prevent ARDS in mice with post-viral acute lung injury.

We will randomize patients with confirmed COVID19 with acute hypoxic respiratory failure (O2 saturation below 93% on minimal 2l/min O2 therapy; and/or PaO2/FiO2 below 350 mmHg) to receive up to 14 days of SC Zilucoplan® on top of standard of care (active group A), or to receive standard of care treatment (control group B). Randomization will be done at a 2:1 ratio active: control group. In the active group A, patients will additionally receive daily antibiotics (daily 3rd generation cephalosporin IV while in hospital, followed by oral ciprofloxacin while discharged) as primary prophylaxis against meningococcal disease until 14 days after the last dose of Zilucoplan®. Control group B will receive standard of care and prophylactic antibiotics (3rd generation cephalosporin IV) for only 1 week (or until hospital discharge whichever comes first), to control for the effects of antibiotics on the clinical course of COVID-19. In case of allergies to these antibiotics, or on clinical indication, these antibiotics may be switched to antibiotics that also cover Neisseria meningitidis.

To measure the effectiveness of Zilucoplan® on restoring lung homeostasis, the primary endpoint of this intervention is measuring change in oxygenation parameters comparing baseline values (pretreatment) to values predose day 6 and to values at day 15 (or discharge whichever comes first) post-randomizationin group A and group B and the differences in these values between group A and group B.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≥6 days and ≤16 days of flu-like symptoms or malaise prior to randomization) infection with COVID-19.
* COVID-19 diagnosis confirmed by antigen detection test and/or PCR and/or positive serology, or any emerging and validated diagnostic laboratory test for COVID-19 within this period. For patients with a negative SARS-CoV-2 PCR and either a positive SARS-CoV-2 antigen or antibody test, the presence of suggestive lesions for COVID-19 on chest-CT scan is mandatory.
* In some patients, it may be impossible to get a confident laboratory confirmation of COVID-19 diagnosis after 24h of hospital admission because viral load is low and/or problems with diagnostic sensitivity. In those cases, in absence of an alternative diagnosis, and with highly suspect bilateral ground glass opacities on recent (<24h) chest-CT scan (confirmed by a radiologist and pulmonary physician as probable COVID-19), and a typical clinical and chemical diagnosis with signs of cytokine release syndrome, a patient can be enrolled as probable SARS-CoV-2-infected. In all cases, this needs confirmation by later seroconversion.
* Presence of hypoxia defined as :

  * O2 saturation below 93% on minimal 2l/min O2 therapy; and/or
  * PaO2/FiO2 below 350 mmHg (Strongly recommended: patient in upright position, after minimal 3 minutes without supplemental oxygen; In ventilated patients or ECMO patients PaO2 can be taken from invasive arterial line and FiO2 taken directly from mechanical ventilation settings).
* Signs of acute lung injury and/or cytokine release syndrome defined as ANY of the following

  * serum ferritin concentration >1000 mcg/L and rising since last 24h
  * single ferritin above 2000 mcg/L in patients requiring immediate high flow oxygen device (Optiflow) or non-invasive or invasive mechanical ventilation
  * lymphopenia defined as <800 lymphocytes/microliter and two of the following extra criteria

    * Ferritin > 700 mcg/L and rising since last 24h
    * Increased LDH (above 300 IU/L) and rising since last 24h
    * D-Dimers > 1000 ng/mL and rising since last 24h
    * CRP above 70 mg/L and rising since last 24h and absence of bacterial infection
    * if three of the above are present at admission, no need to document 24h rise
* Low dose Chest CT or HRCT or Angio Chest CT scan showing bilateral infiltrates within last 2 days prior to randomisation
* Admitted to specialized COVID-19 ward or an ICU ward taking care of COVID-19 patients
* Age ≥ 18 years
* Women of childbearing potential must have a negative serum pregnancy test pre-dose on day 1. Women of childbearing potential must consistently and correctly use (during the entire treatment period and 4weeks after last Zilucoplan® administration ) at least 1 highly effective method for contraception.
* Willing and able to provide informed consent or legal representative willing to provide informed consent

Exclusion Criteria:

* Patients with known history of serious allergic reactions, including anaphylaxis, to Zilucoplan® or inability to receive antibiotic prophylaxis due to allergy to ALL of the antibiotics that can be given for prophylaxis of meningococcal disease
* History of active or past meningococcal disease
* Invasive mechanical ventilation > 24 h at randomization
* Patient on ECMO at screening
* Clinical frailty scale above 3 before onset of the COVID-19 episode
* Weight below 54 kg as measured max 1 week prior to inclusion
* Weight above 150 kg as measured max 1 week prior to inclusion
* Active bacterial or fungal infection
* Unlikely to survive beyond 48h
* Neutrophil count below 1500 cells/microliter
* Platelets below 50.000/microliter
* Patients enrolled in another investigational drug study
* Patients on high dose systemic steroids (> 8 mg methylprednisolone or equivalent for more than 1 month) or other moderately immunosuppressive drugs (in the opinion of the investigator) for COVID19 unrelated disorder
* Patients on current complement inhibiting drugs
* Serum transaminase levels >5 times upper limit of normal, unless there are clear signs of cytokine release syndrome defined by LDH >300 IU/L and ferritin >700 ng/ml
* Pregnant or breastfeeding females (all female subjects deemed of childbearing potential by the investigator must have negative pregnancy test at screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart N Lambrecht, MDPhD, Principal Investigator — University Ghent
Locations (9):
- Belgium (9):
  - OLVZ Aalst, Aalst
  - AZ Sint Jan Brugge, Bruges
  - Erasmus University Hospital, Brussels
  - AZ Sint-Lucas, Ghent
  - University Hospital Ghent, Ghent
  - Jan Yperman Ziekenhuis Ieper, Ieper
  - University Hospital Liège, Liège
  - AZ Delta, Roeselare
  - AZ Vesalius, Tongeren

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Leeuw E, Van Damme KFA, Declercq J, Bosteels C, Maes B, Tavernier SJ, Detalle L, Smart T, Glatt S, Debeuf N, Deckers J, Lameire S, Vandecasteele SJ, De Neve N, Demedts IK, Govaerts E, Knoop C, Vanhove K, Moutschen M, Terryn W, Depuydt P, Van Braeckel E, Haerynck F, Hendrickx TCJ, Parrein V, Lalla M, Brittain C, Lambrecht BN. Efficacy and safety of the investigational complement C5 inhibitor zilucoplan in patients hospitalized with COVID-19: an open-label randomized controlled trial. Respir Res. 2022 Aug 9;23(1):202. doi: 10.1186/s12931-022-02126-2. PMID 35945604
- [Derived] Declercq J, Bosteels C, Van Damme K, De Leeuw E, Maes B, Vandecauter A, Vermeersch S, Delporte A, Demeyere B, Vuylsteke M, Lalla M, Smart T, Detalle L, Bouw R, Streffer J, Degeeter T, Vergotte M, Guisez T, Van Braeckel E, Van Der Straeten C, Lambrecht BN. Zilucoplan in patients with acute hypoxic respiratory failure due to COVID-19 (ZILU-COV): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 19;21(1):934. doi: 10.1186/s13063-020-04884-0. PMID 33213529

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 patients were randomized at the 9 participating centers.
Groups:
- Group A (Active): Standard of Care (SoC) + subcutaneous Zilucoplan® + prophylactic antibiotics until 14 days after last Zilucoplan®
  Zilucoplan®: 14 days of SC Zilucoplan® 32.4mg once daily on top of standard of care + prophylactic antibiotics until 14 days after last Zilucoplan®
- Group B (Control): Standard of Care (SoC) + 1 week of prophylactic antibiotics (or until hospital discharge, whichever comes first)
  Placebo: standard of care treatment + 1 week of prophylactic antibiotics + 1 week of prophylactic antibiotics (or until hospital discharge, whichever comes first)
Period: Overall Study
Arm/Group | Group A (Active) | Group B (Control)
Started (randomized patients) | 55 | 26
Treated (patients that received at least 1 intervention) | 54 | 24
Completed (included in safety and primary analysis) | 54 | 24
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — did not receive allocated intervention due to clinical error | 0 | 1
Not completed — did not meet inclusion criteria but was randomized without receiving the allocated intervention | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Active) | Group B (Control) | Total
Number analyzed (Participants) | 54 | 24 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 12 | 41
  >=65 years | 25 | 12 | 37
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 83] | 64.8 [50 to 85] | 63 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 49 | 19 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 23 | 77
  Unknown or Not Reported | 0 | 1 | 1
Ordinal scale for clinical improvement [Count of Participants; unit: Participants] — 6-point ordinal scale: 1 death, 2 on invasive mechanical ventilation or ECMO (ExtraCorporeal Membrane Oxygenation; 3 on non-invasive ventilation of high flow oxygen devices; 4 hospitalized, requiring supplemental oxygen; 5 hospitalized, not requiring supplemental oxygen, 6 not hospitalized
  Participants
    2. on invasive mechanical ventilation of ECMO | 8 | 2 | 10
    3. on non-invasive ventilation of high flow oxygen devices | 19 | 8 | 27
    4. hospitalized, requiring supplemental oxygen | 26 | 14 | 40
    5. hospitalized, not requiring supplemental oxygen | 1 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  African | 4 | 0 | 4
  Arabian | 3 | 1 | 4
  Asian | 1 | 0 | 1
  Caucasian | 46 | 22 | 68
  Other | 0 | 1 | 1
Sequential Organ Failure Assessment (SOFA score) [Count of Participants; unit: Participants] — The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems (respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). The score is calculated based on the worst values in the previous 24h at time of evaluation. Score ranges from 0 (best) to 24 (worst) points.
  SOFA score 0-1: mortality 0%; SOFA score 2-3: mortality 6.4%; SOFA score 4-5: mortality 20.2%; SOFA score 6-7: mortality 21.5%; SOFA score 8-9: mortality 33.3%; Population: For 4 participants, not all information was present to calculate the SOFA score at baseline.
  Participants
    number analyzed (Participants) | 51 | 23 | 74
    score 1-2 | 29 | 14 | 43
    score 3-4 | 14 | 7 | 21
    score 5-6 | 1 | 2 | 3
    score 7-8 | 7 | 0 | 7
Arterial hypertension [Count of Participants; unit: Participants]
  yes | 26 | 10 | 36
  no | 28 | 14 | 42
Diabetes mellitus [Count of Participants; unit: Participants]
  yes | 26 | 10 | 36
  no | 28 | 14 | 42
Cardiovascular disease [Count of Participants; unit: Participants]
  yes | 9 | 10 | 19
  no | 45 | 14 | 59
Chronic kidney disease [Count of Participants; unit: Participants]
  yes | 4 | 0 | 4
  no | 50 | 24 | 74
Glucocorticoids at randomisation [Count of Participants; unit: Participants]
  yes | 49 | 18 | 67
  no | 5 | 6 | 11
glucocorticoid use during first 28 days [Count of Participants; unit: Participants]
  yes | 52 | 21 | 73
  no | 2 | 3 | 5
Anticoagulants at randomisation [Count of Participants; unit: Participants]
  yes | 49 | 21 | 70
  no | 5 | 3 | 8
Antibiotics at randomisation [Count of Participants; unit: Participants]
  yes | 16 | 2 | 18
  no | 38 | 22 | 60
Remdesivir at randomisation [Count of Participants; unit: Participants]
  yes | 7 | 2 | 9
  no | 47 | 22 | 69
PaO2/FiO2 ratio at baseline [Mean (Standard Deviation); unit: mmHG] | 169.2 (93.8) | 175.1 (92.5) | 171.1 (92.8)
A-a gradient at baseline [Mean (Standard Deviation); unit: mmHg] | 271.8 (211.1) | 237.2 (207.8) | 260.6 (209.2)
Days of hospitalization at randomisation [Median (Full Range); unit: days] | 3 [1 to 8] | 2 [1 to 11] | 2 [1 to 11]
Days of symptoms at randomisation [Median (Full Range); unit: days] | 10 [7 to 16] | 10 [6 to 13] | 10 [6 to 16]
Admitted to ICU at randomisation [Count of Participants; unit: Participants] | 30 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygenation
Description: defined by Pa02/FiO2 ratio while breathing room air, P(Aa)O2 gradient and a/A pO2 ratio
Time Frame: at predose, day 6 and day 15 (or at discharge, whichever comes first)
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 52 | 20
mmHg
  change from baseline in PaO2/FiO2 day 6 | 56.4 [31.9 to 80.9] | 20.6 [17.3 to 58.5]
  change from baseline in PaO2/FiO2 day 15 | 123.5 [94.3 to 152.7] | 83.7 [39.0 to 128.4]
  change from baseline in a/A PO2 day 6 | 0.10 [0.06 to 0.15] | 0.04 [0.04 to 0.11]
  change from baseline in a/A PO2 day 15 | 0.25 [0.19 to 0.31] | 0.17 [0.08 to 0.26]

2. Primary Outcome: Change in Oxygenation
Description: defined by Pa02/FiO2 ratio while breathing room air, P(Aa)O2 gradient and a/A pO2 ratio
Time Frame: at predose, day 6 and day 15 (or at discharge, whichever comes first)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 52 | 20
mmHg
  (A-a) gradient day 6 | 114.6 [92.6 to 141.9] | 146.7 [105.4 to 204.3]
  (A-a) gradient day 15 | 58.6 [44.9 to 76.5] | 86.9 [57.9 to 130.6]

3. Secondary Outcome: Mean Change in 6-point Ordinal Scale Change for Clinical Improvement
Description: 6-point ordinal scale defined as
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Not hospitalized
Time Frame: between day 1 and respectively day 6, day 15 (or discharge, whichever comes first) and day 28 (by phone call).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
score on a scale
  mean change in 6-point ordinal scale change day 6 | 0.1 (1.0) | 0.1 (0.9)
  mean change in 6-point ordinal scale change day 15 | 1.2 (1.4) | 1 (1.5)
  mean change in 6-point ordinal scale change day 28 | 1.7 (1.5) | 1.3 (1.8)

4. Secondary Outcome: Number of Days With Hypoxia
Description: defined as SpO2 < 93% breathing room air or the dependence on supplemental oxygen
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 13 [3 to 28] | 10 [2 to 28]

5. Secondary Outcome: Number of Days of Supplemental Oxygen Use
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 13 [3 to 28] | 10 [2 to 28]

6. Secondary Outcome: Time to Absence of Fever (Defined as 37.1°C or More) for More Than 48h Without Antipyretic
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 7 [1 to 28] | 3 [1 to 28]

7. Secondary Outcome: Number of Days With Fever
Description: defined as 37.1°C or more
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 7 [0 to 28] | 4 [0 to 20]

8. Secondary Outcome: Mean Change in CRP Levels Between Day 1 and Day 6
Time Frame: day 1, day 6
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
mg/mL | -89.6 (91.5) | -100 (61.9)

9. Secondary Outcome: Mean Change in CRP Levels Between Day 1 and Day 15 (or Discharge Whichever Comes First)
Time Frame: day 1, day 15
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
mg/mL | -91.0 (106.3) | -96.2 (98.4)

10. Secondary Outcome: Mean Change in Ferritin Levels Between Day 1 and Day 6
Time Frame: day 1, day 6
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
µg/L | -544.4 (1489.9) | -282.3 (517.0)

11. Secondary Outcome: Mean Change in Ferritin Levels Between Day 1 and Day 15 (or Discharge, Whichever Comes First)
Time Frame: day 1, day 15
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
µg/L | -201.0 (6204.5) | -303.9 (948.4)

12. Secondary Outcome: Number of Participants With Adverse Events
Description: Any untoward medical occurrence in a subject to whom a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: during hospital admission (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 39 | 17

13. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event is any untoward medical occurrence that:
  * results in death
  * is life-threatening
  * requires inpatient hospitalisation or prolongation of existing hospitalisation
  * results in persistent or significant disability/incapacity
  * consists of a congenital anomaly or birth defect Other 'important medical events' may also be considered serious if they jeopardise the subject or require an intervention to prevent one of the above consequences.
  NOTE: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.
Time Frame: at 10-20 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 10 | 5

14. Secondary Outcome: Number of Participants With SUSAR's (Suspected Unexpected Serious Adverse Reaction)
Description: A serious adverse reaction, the nature and severity of which is not consistent with the information about the medicinal product in question set out:
  * in the case of a product with a marketing authorisation, in the summary of product characteristics (SmPC) for that product
  * in the case of any other investigational medicinal product, in the investigator's brochure (IB) relating to the study in question
Time Frame: during hospital admission (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With SAR's (Serious Adverse Reaction)
Description: An adverse event that is both serious and, in the opinion of the reporting Investigator, believed with reasonable probability to be due to one of the study treatments, based on the information provided.
Time Frame: during hospital admission (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 0 | 0

16. Secondary Outcome: Duration of Hospital Stay
Time Frame: at 12-22 weeks follow-up
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 15 [5 to 74] | 13 [3 to 43]

17. Secondary Outcome: Duration of Hospital Stay in Survivors
Time Frame: at 12-22 weeks follow-up
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 47 | 19
days | 15 [5 to 74] | 12 [3 to 43]

18. Secondary Outcome: Number of Participants With Improvement, No Change, Death or Deterioration in SOFA Score Between Day 1 and Day 6 (or on Discharge, Whichever is First)
Description: The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems (respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). Score ranges from 0 (best) to 24 (worst) points.
Time Frame: day 1, day 6 or on discharge, whichever is first
Population: Change of SOFA score between day 1 and day 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 43 | 21
Participants
  improvement or discharge | 21 | 10
  no change | 11 | 6
  death or deterioration | 11 | 5

19. Secondary Outcome: Number of Participants With Improvement, No Change, Death or Deterioration in SOFA Score Between Day 1 and Day 15 (or on Discharge, Whichever is First)
Description: as for outcome 18
Time Frame: day 1, day 15 or on discharge, whichever is first
Population: Change of SOFA score between day 1 and day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 43 | 17
Participants
  improvement or discharge | 33 | 12
  no change | 5 | 1
  death or deterioration | 5 | 4

20. Secondary Outcome: Number of Participants With Nosocomial Bacterial or Invasive Fungal Infection for 28 Days (Phone Call) After Enrollment in Trial
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 12 | 4

21. Secondary Outcome: Median Time to at Least a 2-point Improvement on the 6-point Ordinal Scale or Discharge During the 28-day Assessment Period (Range) - Days
Description: The 6-point ordinal scale for clinical improvement is defined as 1 = Death; 2 = Hospitalized, on invasive mechanical ventilation or ECMO; 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4 = Hospitalized, requiring supplemental oxygen; 5 = Hospitalized, not requiring supplemental oxygen; 6 = Not hospitalized. A higher score represent a better outcome
Time Frame: Day 28
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 15 [2 to 28] | 12 [6 to 28]

22. Secondary Outcome: Number of Participants in Each Category of the 6- Point Ordinal Scale for Clinical Improvement
Description: as for outcome 21
Time Frame: at 12-22 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 44 | 19
Participants
  category 2 | 0 | 0
  category 3 | 0 | 0
  category 4 | 1 | 0
  category 5 | 0 | 0
  category 6 | 43 | 19

23. Secondary Outcome: Number of Participants in Each Category of the WHO Performance Scale
Description: The WHO performance status classification categorises patients as:
  0: able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. symptomatic and in a chair or in bed for greater than 50% of the day but not bedridden
  4. completely disabled; cannot carry out any self-care; totally confined to bed or chair.
Time Frame: during hospital admission (up to 28 days)
Population: For 1 participant of group A and 1 participant of group B, the WHO performance scale was not recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 43 | 18
Participants
  category 0 | 23 | 10
  category 1 | 18 | 7
  category >=2 | 2 | 1

24. Secondary Outcome: Result of 6 Minute Walk Test
Description: Distance in 6 minute walk test. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. Total distance in meters. A higher score has a better outcome
Time Frame: at 12-22 weeks follow-up
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
meters | 539.7 (107.7) | 490.6 (0.18)

25. Secondary Outcome: All-cause Mortality Rate (Excluding Group That Entered During Ventilation)
Time Frame: at day 28
Population: Population excluding patients that required invasive mechanical ventilation or ECMO within 24 hours prior to or after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 45 | 22
Participants | 3 | 5

26. Secondary Outcome: All-cause Mortality Rate (Including Group That Entered During Ventilation)
Time Frame: at day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 5 | 5

27. Secondary Outcome: All Cause Mortality for the Entire Study Population
Time Frame: at follow up 12-22 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 7 | 5

28. Other Pre Specified Outcome: Number of Ventilator-free Days
Time Frame: day 1, day 28 or discharge whichever comes first
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 7 [0 to 27] | 9 [0 to 28]

29. Other Pre Specified Outcome: Time Since Randomization to Progression to ARDS (Acute Respiratory Distress Syndrome)
Description: criteria-defined ARDS criteria-defined ARDS according to the adapted Berlin criteria as follow:
  * within 1 week of a known Clinical insult or new or worsening respiratory symptoms
  * bilateral infiltrates not supposed to be of cardiac origin or fluid overload
  * PaO2/FiO2 < 300 mmHg
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 1 [1 to 14] | 3 [1 to 10]

30. Other Pre Specified Outcome: Number of Participants With Lung Fibrosis on Chest CT Scan at Follow up
Time Frame: at 12-22 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
Participants | 0 | 0

31. Other Pre Specified Outcome: Time Since Randomization Until Improvement in Oxygenation
Description: defined as independence from supplemental oxygen
Time Frame: during hospital admission (up to 28 days)
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) | Group B (Control)
Number analyzed (Participants) | 54 | 24
days | 13 [3 to 28] | 10 [2 to 28]

ADVERSE EVENTS:
Time Frame: All-cause mortality monitored for up to 22 weeks, serious adverse events monitored for up to 20 weeks and other adverse events monitored for up to 28 days.
Description: Some patients encountered several (serious) adverse events. Therefore, the total count of (serious) adverse events can be higher than the number of affected participants.
Arm/Group | Group A (Active) | Group B (Control)
All-Cause Mortality (participants affected / at risk) | 7/54 | 5/24
Serious Adverse Events (participants affected / at risk) | 10/54 | 5/24
Other Adverse Events (participants affected / at risk) | 39/54 | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Active) (N=54) | Group B (Control) (N=24)
Cardiac arrest (Cardiac disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Aspergillus infection (Immune system disorders) | 1 | 0
hypoxic-sichaemic encephalopathy (Nervous system disorders) | 0 | 1
death (General disorders) | 1 | 0
multiple organ dysfunction syndrome (General disorders) | 1 | 0
acute kidney injury (Renal and urinary disorders) | 1 | 1
thrombosis in device (Product Issues) | 0 | 1
bronchopulmonary aspergillus (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
covid-19 (Infections and infestations) | 1 | 0
cytomegalovirus infection (Infections and infestations) | 1 | 0
enterococcal sepsis (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 1 | 0
sepsis (Infections and infestations) | 1 | 0
septic shock (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Active) (N=54) | Group B (Control) (N=24)
hypertension (Vascular disorders) | 8 | 2
alanine animontransferase increased (Investigations) | 4 | 1
aspartate animontransferase increased (Investigations) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
pneumonia pseudomonal (Respiratory, thoracic and mediastinal disorders) | 0 | 2
anemia (Blood and lymphatic system disorders) | 4 | 2
anxiety (Psychiatric disorders) | 6 | 1
delirium (Psychiatric disorders) | 3 | 1
insomnia (Psychiatric disorders) | 5 | 0
constipation (Gastrointestinal disorders) | 7 | 5
decreased appetite (Metabolism and nutrition disorders) | 1 | 2
hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
hypoalbuminia (Metabolism and nutrition disorders) | 3 | 0
pneumonia (Infections and infestations) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04382755/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04382755/SAP_001.pdf